CLINICAL TRIAL: NCT03139006
Title: Diagnostic Accuracy of Spectral Computed Tomography for Detection of Flow Limiting Coronary Stenosis Using Fractional Flow Reserve as the Standard of Reference
Brief Title: Application of speCtraL Computed tomogrAphy to impRove specIficity of Cardiac compuTed tomographY
Acronym: CLARITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Tim Leiner, Prof. Dr., UMC Utrecht
Other Study IDs: NL55917.041.16
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Coronary Stenosis; Myocardial Ischemia; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Stenosis; Myocardial Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Dual-layer spectral detector CT — A dual energy CT approach
  Other Names: SDCT

SUMMARY:
Cardiovascular disease remains the leading cause of morbidity and mortality worldwide. Coronary computed tomography angiography (CCTA) and, if indicated, invasively measured fractional flow reserve (FFR) is currently used for ruling out significant coronary artery disease. FFRCT is a novel non-invasive technique in which FFR is derived from CT images, however this method is currently, just like CCTA, lacking specificity. Spectral Detector CT (SDCT) is a novel technique whereby a spectrum of monoenergetic images at different kiloelectron Volt (keV) values (40 to 200 keV) can be reconstructed. By using these monoenergetic images, a decrease in blooming and beam-hardening artifacts could be achieved. In addition, SDCT offers the opportunity to assess myocardial iodine distribution and quantification. When combining these factors, we hypothesize more accurate information will be available about the coronary anatomy, degree of stenosis and FFRCT and thereby contribute to a more accurate way for the detection of hemodynamic significant stenosis. Therefore, the aim of this study is to assess the accuracy of SDCT as a non-invasive way for the detection of hemodynamically significant coronary artery stenosis.

Objective: The overall objective of this project is to assess the accuracy of SDCT for the detection of flow limiting stenosis in the coronary arteries using invasive FFR as the standard of reference. Whereby different sub-aims (e.g. improvement of FFRCT) are made to answer the overall objective. The secondary objective is to determine the decrease of calcium blooming of calcifications and beam-hardening artifacts and the improvement of myocardial blood volume quantification on SDCT in comparison with conventional CT.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Suspected or known stable angina with pre-test likelihood of 50-85% for obstructive coronary disease, using the method recommended by the European Society of Cardiology 2013 Guidelines on the management of stable coronary artery disease (Eur Heart J 2013);
* Referred for invasive testing with fractional flow reserve;
* Willing and able to give informed consent. The consent procedures, as set by the Institutional Review Board (IRB) will be followed.

Exclusion Criteria:

* Subjects with suspected or known stable angina with pre-test likelihood of 0-50% using the method recommended by the European Society of Cardiology 2013 Guidelines on the management of stable coronary artery disease (Eur Heart J 2013 [24]);
* Subjects who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent or tolerate the coronary CTA examination;
* Subjects with (severe) renal insufficiency, indicated as glomerular filtration rate (GFR) <60 ml/min;
* Subjects with unknown GFR or obtained >3 months before the planned scan;
* Contraindication or allergy to intravenous contrast agent(s);
* Subjects who participate in an other study with radiation which is estimated to be in risk category III (ICRP 62);
* Subjects who are pregnant;
* Subjects with contraindications to cardiac CT and/or S&S protocol, intravenous contrast, intravenous adenosine, betablockers or nitroglycerine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants ≥18 years of age with suspected or known stable angina with pre-test likelihood of 50-85% for obstructive coronary disease (Eur Heart J 2013 guidelines on stable CAD) and who are referred for clinical invasive FFR.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2021-03-29 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Flow limiting stenosis in the coronary arteries defined by invasive fractional flow reserve (FFR) | within 30 days
  An invasive FFR <0.8 indicates a flow limiting stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Tim Leiner, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center UtrechtU, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Hamersvelt RW, Isgum I, de Jong PA, Cramer MJM, Leenders GEH, Willemink MJ, Voskuil M, Leiner T. Application of speCtraL computed tomogrAphy to impRove specIficity of cardiac compuTed tomographY (CLARITY study): rationale and design. BMJ Open. 2019 Mar 1;9(3):e025793. doi: 10.1136/bmjopen-2018-025793. PMID 30826767